CLINICAL TRIAL: NCT00058240
Title: A Dose-Escalation Study of Flavopiridol (NSC 649890) Administered as a 30 Minute Loading Dose Followed by a 4-Hour Infusion in Patients With Previously Treated B-Cell Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)
Brief Title: Flavopiridol in Treating Patients With Previously Treated Chronic Lymphocytic Leukemia or Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01435; NCI-2012-01435 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000287197; NCI-5746; OSU-0055; OSU 0055 (Other: Ohio State University Medical Center); 5746 (Other: CTEP); R21CA112947 (NIH); P30CA016058 (NIH); U01CA076576 (NIH)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — alvocidib

ARMS (1):
- Arm I (Experimental): Patients receive a loading dose of flavopiridol IV over 30 minutes followed by a 4-hour infusion on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for up to 6 courses in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: alvocidib

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275

SUMMARY:
This phase I/II trial studies the side effects and best dose of flavopiridol in treating patients with previously treated chronic lymphocytic leukemia or lymphocytic lymphoma. Drugs used in chemotherapy such as flavopiridol work in different ways to stop cancer cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicity profile, dose-limiting toxicity, and maximum tolerated dose of flavopiridol administered as a 30 minute loading dose followed by a 4-hour infusion once weekly for 4 consecutive weeks every 6 weeks.

II. To determine the safety and feasibility of performing dose escalation to 80 mg/m2 (30 mg/m2 30-minute IV bolus followed by 50 mg/m2 4-hour IV infusion) beginning dose 2 in patients who do not experience severe tumor lysis requiring hemodialysis during dose 1.

III. To determine the pharmacokinetics and cellular pharmacodynamics of flavopiridol administered in this schedule.

SECONDARY OBJECTIVES:

I. To determine the complete response (CR) and overall response rate (CR + PR) of flavopiridol in patients with previously-treated CLL administered as a 30 minute loading dose followed by a 4 hour infusion once weekly for 4 consecutive weeks every 6 weeks.

OUTLINE: This is a dose-escalation study.

Patients receive a loading dose of flavopiridol IV over 30 minutes followed by a 4-hour infusion on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for up to 6 courses in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. After the MTD is determined, 12 additional patients are accrued and treated as above at the recommended phase II dose.

After completion of study treatment, patients are followed at 2 months and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B-cell chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma, including Waldenstrom's macroglobulinemia, as indicated by the following:

  * Massive or progressive splenomegaly and/or lymphadenopathy
  * Anemia (hemoglobin less than 11 g/dL) or thrombocytopenia (platelet count less than 100,000/mm^3)
  * Weight loss of more than 10% within the past 6 months
  * Grade 2 or 3 fatigue
  * Fevers greater than 100.5º C or night sweats for more than 2 weeks with no evidence of infection
  * Progressive lymphocytosis with an increase of more than 50% over a 2-month period or anticipated doubling time of less than 6 months
* Received at least 1 prior therapy for CLL
* Performance status - ECOG (Eastern Cooperative Oncology Group) 0-2
* See Disease Characteristics
* WBC (white blood count) less than 200,000/mm^3
* Bilirubin no greater than 1.5 times normal (unless due to Gilbert's disease or any of the conditions stated below)*
* AST (aspartate aminotransferase) no greater than 2 times normal*
* Creatinine no greater than 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy that would limit survival to less than 2 years
* No history of inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis) unless inactive for more than 2 years
* No psychiatric condition that would preclude compliance with treatment or giving informed consent
* No other concurrent chemotherapy
* No concurrent chronic corticosteroids
* No concurrent hormonal therapy except steroids for new adrenal failure or hormonal agents for nondisease-related conditions (e.g., insulin for diabetes)
* No concurrent dexamethasone or other corticosteroid-based antiemetics
* No concurrent radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-04 (Actual); Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Byrd, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Ni W, Ji J, Dai Z, Papp A, Johnson AJ, Ahn S, Farley KL, Lin TS, Dalton JT, Li X, Jarjoura D, Byrd JC, Sadee W, Grever MR, Phelps MA. Flavopiridol pharmacogenetics: clinical and functional evidence for the role of SLCO1B1/OATP1B1 in flavopiridol disposition. PLoS One. 2010 Nov 1;5(11):e13792. doi: 10.1371/journal.pone.0013792. PMID 21072184
- [Result] Pierceall WE, Warner SL, Lena RJ, Doykan C, Blake N, Elashoff M, Hoff DV, Bearss DJ, Cardone MH, Andritsos L, Byrd JC, Lanasa MC, Grever MR, Johnson AJ. Mitochondrial priming of chronic lymphocytic leukemia patients associates Bcl-xL dependence with alvocidib response. Leukemia. 2014 Nov;28(11):2251-4. doi: 10.1038/leu.2014.206. Epub 2014 Jul 3. No abstract available. PMID 24990615
- [Result] Lin TS, Ruppert AS, Johnson AJ, Fischer B, Heerema NA, Andritsos LA, Blum KA, Flynn JM, Jones JA, Hu W, Moran ME, Mitchell SM, Smith LL, Wagner AJ, Raymond CA, Schaaf LJ, Phelps MA, Villalona-Calero MA, Grever MR, Byrd JC. Phase II study of flavopiridol in relapsed chronic lymphocytic leukemia demonstrating high response rates in genetically high-risk disease. J Clin Oncol. 2009 Dec 10;27(35):6012-8. doi: 10.1200/JCO.2009.22.6944. Epub 2009 Oct 13. PMID 19826119
- [Result] Woyach JA, Lozanski G, Ruppert AS, Lozanski A, Blum KA, Jones JA, Flynn JM, Johnson AJ, Grever MR, Heerema NA, Byrd JC. Outcome of patients with relapsed or refractory chronic lymphocytic leukemia treated with flavopiridol: impact of genetic features. Leukemia. 2012 Jun;26(6):1442-4. doi: 10.1038/leu.2011.375. Epub 2012 Jan 13. No abstract available. PMID 22289993

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with relapsed, symptomatic Chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) were enrolled and received treatment between May 2003 and February 2006
Groups:
- Dose Level 1: Patients were administered Flavopiridol 30mg/m2 bolus followed by 30 mg/m2 4 hour infusion weekly for four weeks followed by two weeks without therapy for a total of 6 cycles
- Dose Level 2: Patients were administered Flavopiridol 40mg/m2 bolus followed by 40 mg/m2 4 hour infusion weekly for four weeks followed by two weeks without therapy for a total of 6 cycles
- Dose Level 3: Patients were administered Flavopiridol dose level one scheduled for the first cycle. In absence of severe toxicity, dose level was escalated to 30mg/m2 bolus followed by 50 mg/m2 4 hour infusion for a total of 6 cycles
- Dose Level 4: Patients were administered Flavopiridol dose level one scheduled for the first dose. In absence of severe toxicity, dose level was escalated to 30mg/m2 bolus followed by 50 mg/m2 4 hour infusion for a total of 6 cycles
Period: First Dose Level
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Started | 20 | 3 | 17 | 12
Treated | 20 | 3 | 17 | 12
Completed | 20 | 3 | 17 | 12
Not Completed | 0 | 0 | 0 | 0
Period: Second Dose Level
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Started | 0 | 0 | 2 (2 patients were previously treated at Dose level 1, relapsed, and retreated at Dose level 3.) | 4 (4 patients previously relapsed on a different Dose level and were retreated at Dose level 4.)
Completed | 0 | 0 | 2 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 52 unique patients due to 6 patients being
Groups:
- Dose Level 1: Dose Level 1: Patients were administered Flavopiridol 30mg/m2 bolus followed by 30 mg/m2 4 hour infusion weekly for four weeks followed by two weeks without therapy for a total of 6 cycles
- Dose Level 2: Dose Level 2: Patients were administered Flavopiridol 40mg/m2 bolus followed by 40 mg/m2 4 hour infusion weekly for four weeks followed by two weeks without therapy for a total of 6 cycles.
- Dose Level 3: Dose Level 3: Patients were administered Flavopiridol dose level one scheduled for the first cycle. In absence of severe toxicity, dose level was escalated to 30mg/m2 bolus followed by 50 mg/m2 4 hour infusion for a total of 6 cycles
- Dose Level 4: Dose Level 4: Patients were administered Flavopiridol dose level one scheduled for the first dose. In absence of severe toxicity, dose level was escalated to 30mg/m2 bolus followed by 50 mg/m2 4 hour infusion for a total of 6 cycles
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Total
Number analyzed (Participants) | 20 | 3 | 17 | 12 | 52
Age, Continuous [Median (Full Range); unit: years] | 61.5 [44 to 84] | 52 [44 to 62] | 55 [39 to 69] | 60 [38 to 75] | 60 [38 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 3 | 3 | 14
  Male | 14 | 1 | 14 | 9 | 38
Region of Enrollment [Number; unit: patients]
  United States | 20 | 3 | 17 | 12 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicities (DLTs)
Description: DLTs were defined as non-hematologic toxicity of grade 3 or greater severity (excluding transient liver function abnormalities, transient electrolyte abnormalities that are not life threatening, fatigue, or diarrhea that resolve within 4 days), or in some case grade 2 toxicity (i.e. irreversible renal, chronic pulmonary, neurologic, or cardiac toxicity). Hematologic toxicity were evaluated by the modified NCI criteria and followed closely. Dose limiting only if grade 4 thrombocytopenia or neutropenia persists for 7 days or greater. Inability to continue with cycle 2 by 7 weeks for reasons other than progression of disease will also be considered a DLT.The National Cancer Institute Common Toxicity Criteria will be used to characterize toxicity.
Time Frame: up to 7 weeks
Measure: Number; unit: patients
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 20 | 3 | 19 | 16
patients | 2 | 2 | 4 | 3

2. Primary Outcome: Recommended Dose Level of Flavopiridol
Description: Recommended dose determined by number of DLTs [non-hematologic toxicity grade 3 or greater (excluding not life-threatening transient liver function or transient electrolyte abnormalities, fatigue, or diarrhea resolving within 4 days), some grade 2 toxicity (i.e. irreversible renal, chronic pulmonary, neurologic, or cardiac toxicity), hematologic toxicity of grade 4 thrombocytopenia/neutropenia persisting for 7 days or greater, or inability to continue cycle 2 by 7 weeks for reasons other than disease progression] and consideration of number of patients with severe tumor lysis requiring hemodialysis with dose 1.
Time Frame: Up to 6 weeks
Measure: Number; unit: mg/m^2
Groups:
- Dose Level 4: Flavopiridol was escalated to 30mg/m2 bolus followed by 50 mg/m2 4 hour beginning Dose Level 2 Cycle 1 for 6 Cycles.
Arm/Group | Dose Level 4
Number analyzed (Participants) | 16
mg/m^2
  Cycle 1 dose 1 | 30
  Cycle 1 dose 2 thru Cycle 6 | 50

3. Secondary Outcome: Overall Response Rate (CR + PR) of Flavopiridol in Patients Evaluated Utilizing the Revised National Cancer Institute-sponsored Working Group Guidelines
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 2 years
Measure: Number; unit: patients
Groups:
- Dose Level 1, 2, 3, 4: Dose Level 1: Patients were administered Flavopiridol 30mg/m2 bolus followed by 30 mg/m2 4 hour infusion weekly for four weeks followed by two weeks without therapy for a total of 6 cycles Dose Level 2: Patients were administered Flavopiridol 40mg/m2 bolus followed by 40 mg/m2 4 hour infusion weekly for four weeks followed by two weeks without therapy for a total of 6 cycles.
  Dose Level 3: Patients were administered Flavopiridol dose level one scheduled for the first cycle. In absence of severe toxicity, dose level was escalated to 30mg/m2 bolus followed by 50 mg/m2 4 hour infusion for a total of 6 cycles Dose Level 4: Patients were administered Flavopiridol dose level one scheduled for the first dose. In absence of severe toxicity, dose level was escalated to 30mg/m2 bolus followed by 50 mg/m2 4 hour infusion for a total of 6 cycles
Arm/Group | Dose Level 1, 2, 3, 4
Number analyzed (Participants) | 52
patients | 21

ADVERSE EVENTS:
Time Frame: Patients were assessed for toxicities from Day 1 of each Flavopiridol Treatment to Post-Treatment Follow-up. Follow up was performed every 3 months for 2 years.
Description: Adverse events were reported for 40 unique patients treated at dose levels 1-3 and 16 patients treated at Dose level 4
Groups:
- Dose Levels 1-3: Dose Level 1: Patients were administered Flavopiridol 30mg/m2 bolus followed by 30 mg/m2 4 hour infusion weekly for four weeks followed by two weeks without therapy for a total of 6 cycles
  Dose Level 2: Patients were administered Flavopiridol 40mg/m2 bolus followed by 40 mg/m2 4 hour infusion weekly for four weeks followed by two weeks without therapy for a total of 6 cycles
  Dose Level 3: Patients were administered Flavopiridol dose level one scheduled for the first cycle. In absence of severe toxicity, dose level was escalated to 30mg/m2 bolus followed by 50 mg/m2 4 hour infusion for a total of 6 cycles
Arm/Group | Dose Levels 1-3 | Dose Level 4
Serious Adverse Events (participants affected / at risk) | 11/42 | 1/16
Other Adverse Events (participants affected / at risk) | 40/40 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Levels 1-3 (N=42) | Dose Level 4 (N=16)
Hyperacute Tumor Lysis (Metabolism and nutrition disorders) | 11 (11) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Levels 1-3 (N=40) | Dose Level 4 (N=16)
Absolute Neutrophil Count (Investigations) | 30 (30) | 16 (16)
WBC (Investigations) | 0 (0) | 11 (11)
Platelets (Investigations) | 15 (15) | 7 (7)
Hemorhage (Vascular disorders) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 16 (16) | 12 (12)
Abdominal pain/cramping (Gastrointestinal disorders) | 2 (2) | 1 (1)
AST SGOT(serum glutamic oxaloacetic transaminase) or ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 13 (13) | 3 (3)
Bilirubin (Investigations) | 3 (3) | 1 (1)
Renal Failture (Renal and urinary disorders) | 1 (1) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Infection w/neutropenia (Infections and infestations) | 7 (7) | 6 (6)
Fatigue (General disorders) | 8 (8) | 2 (2)
Biochemical tumor lysis (Metabolism and nutrition disorders) | 23 (23) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less